CLINICAL TRIAL: NCT02407782
Title: Oral Ivermectin Versus Topical Permethrin to Treat Scabies in Children and Adults: a Cluster Multicenter Randomized Trial
Brief Title: Oral Ivermectin Versus Topical Permethrin to Treat Scabies in Children and Adults
Acronym: SCRATCH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHUBX 2011/16
Record Dates: First submitted 2015-03-24; First posted 2015-04-03 (Estimated); Last update posted 2024-06-17 (Actual); Status verified 2016-06

CONDITIONS: Scabies
Keywords: Scabies; children; cluster; permethrin; Ivermectin; adults
MeSH Terms: conditions — Scabies | interventions — Ivermectin; Permethrin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ivermectin (Experimental)
  Interventions: Drug: Ivermectin
- Permethrin (Experimental)
  Interventions: Drug: Permethrin

INTERVENTIONS:
Drug: Ivermectin — oral ivermectin, 200μg/kg given at baseline and at day 10.
  Arms: Ivermectin
Drug: Permethrin — topical permethrin 5% cream applied at baseline and at day 10.
  Arms: Permethrin

SUMMARY:
Scabies remains a frequent condition that affects adults and children. The aim of this study is to compare the efficacy and safety of two drug treatments against scabies in children and their close contacts. One group will apply topical permethrin 5% and the other group will receive oral ivermectin.

Both groups will be treated twice, once at inclusion and the second time 10 days later. Both treatment regimens have been used widely and are safe to use.

DETAILED DESCRIPTION:
Scabies is a common condition, even in European countries, and the annual incidence seems to have increased over the past several years.

Children and infants represent one-third of patients with scabies. Diagnostic features comprise pruritus, skin burrows and the delta jet wing dermoscopic sign.

In many countries, topical permethrin is the first line therapy. Moreover, oral treatment with ivermectin represents an interesting alternative therapy, usually used as one dose of 200μg/kg, and more and more frequently recommended as two doses (one on day 1 and one between day 8 and day 15) without strong evidence. Management of scabies requires giving a treatment not only to the patient but also to the patient's close contacts.

The objective of our study is to compare efficacy and safety of topical permethrin applied twice at day 1 and day 10 versus oral ivermectin given twice at day 1 and day 10 to treat scabies in children and their close contacts. Children (2 to15 years) with scabies and their close contacts - or first circle- will be randomized 1:1 to receive permethrin or ivermectin.

A clinical follow-up will be performed 28 days (V2) and 56 days (V3) after the inclusion, including a dermatological examination and to collect safety data.

ELIGIBILITY:
Inclusion Criteria:

* children or adult
* For children, weight more than 15 kg
* Documented diagnosis of scabies, defined by positive dermoscopic examination.

Exclusion Criteria:

* Previous scabies therapy during the past 4 weeks
* Known allergy to ivermectin or permethrin
* Widespread eczematization or impetiginization
* Liver or renal failure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1092 (Actual)
Dates: Start 2016-01-19 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
Assessment of skin lesions and healing at day 28 | Day 28
  Healing of skin lesions and disappearance of pruritus at day 28 of the treatment in the cluster composed by the child and its close contacts

SECONDARY OUTCOMES:
Assessment of skin lesions and healing at day 56 | day 56
  Healing of skin lesions and disappearance of pruritus at day 56 of the treatment in the cluster composed by the child and its close contacts.
Assessment of skin lesions and healing at day 28 and 56 in children | Day 28 and Day 56
  Healing of skin lesions and disappearance of pruritus at day 28 and day 56 of the treatment in children
Number of unaffected members in clusters treated by permethrin versus ivermectin at D0, D28 and D56. | day 0, day 28 and d56
Evaluation of delta wing jet sign(s) and mite egs | Day 56
Incidence of serious adverse events | Day 56
  Safety in both groups
adherence of patients | Day 56
  Preference and adherence of patients in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Bruneau Giraudeau, Doctor, Study Chair — Centre d'investigation clinique Inserm 1415 CHRU de Tours
Locations (29):
- France (28):
  - CHU de Bordeaux Hôpital Pellegrin, Bordeaux, Aquitaine
  - CHU de Lyon, Bron, Auvergne-Rhône-Alpes
  - CHG de Chalon sur Saône, Chalon-sur-Saône, Bourgogne-Franche-Comté
  - CHU de Dijon, Dijon, Bourgogne-Franche-Comté
  - CHU de Rennes, Rennes, Brittany Region
  - CHRU de Tours, Tours, Centre-Val de Loire
  - CHU de Montpellier, Montpellier, Languedoc-Roussillon
  - CHU de la Réunion, Saint-Pierre, Martinique
  - CHU d'Angers, Angers, Pays de la Loire Region
  - CH du Mans, Le Mans, Pays de la Loire Region
  - CHU de Nantes, Nantes, Pays de la Loire Region
  - CHI de Fréjus, Fréjus, Provence-Alpes-Côte d'Azur Region
  - CHU de Nice, Nice, Provence-Alpes-Côte d'Azur Region
  - APHP- Bobigny - Avicenne, Bobigny
  - CHU de Bordeaux - Saint André, Bordeaux
  - CHU de Brest, Brest
  - CHD Vendée, La Roche-sur-Yon
  - CH Le Havre, Le Havre
  - CHRU de Lille, Lille
  - AP-HM, Marseille
  - APHP Hôpital Cochin, Paris
  - CH de Périgueux, Périgueux
  - CHU de Reims, Reims
  - CHU de Rouen, Rouen
  - CHU de Saint-Etienne, Saint-Etienne
  - CH d'Argenteuil, Argenteuil, Île-de-France Region
  - CHU de Créteil - Hôpital Henry Mondor, Créteil, Île-de-France Region
  - AP-HP - Hôpital Robert Debré, Paris, Île-de-France Region
- CHU de Pointe à Pitre, Pointe-à-Pitre, Guadeloupe

REFERENCES:
- [Derived] Boralevi F, Simon G, Bernigaud C, Brun J, Goujon E, Perrot JL, Phan A, Herisse AL, Maruani A, Vanhaecke C, Couty E, Abasq-Thomas C, Fournet M, Mallet S, Brenaut E, Hubiche T, Balguerie X, Caux F, Beneton N, Dutkiewicz AS, Adamski H, Aubert H, Bourrat E, Couzan C, Eyraud A, Janela-Lapert R, Marti A, Miquel J, Richard M, Barbarot S, Bonniaud B, Chabbert C, Delion F, Dinulescu M, Duong TA, Etienne M, Hirsch G, Isnard C, Huet F, Le Bidre E, Leducq S, Legrand A, Monestier S, Morice-Picard F, Seneschal J, Capelli A, Lacoste C, Labreze C, Miraglia G, Do-Pham G, Giraudeau B, Chosidow O. Oral ivermectin versus 5% permethrin cream to treat children and adults with classic scabies: multicentre, assessor blinded, cluster randomised clinical trial. BMJ. 2026 Jan 6;392:e086277. doi: 10.1136/bmj-2025-086277. PMID 41494769